CLINICAL TRIAL: NCT05353803
Title: Smart and Healthy Ageing Through People Engaging in Supportive Systems (SHAPES) Digital App and Platform for Supporting Medicines Control and Optimization in Older Individuals With Heart Failure
Brief Title: Digital App and Platform for Supporting Medicines Control and Optimization in Older Individuals With Heart Failure
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Clinika de Kay SL (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Supportive Care
Other Study IDs: UC-PT3-001-CH
Record Dates: First submitted 2022-04-11; First posted 2022-04-29 (Actual); Last update posted 2024-02-08 (Actual); Status verified 2023-08

CONDITIONS: Heart Failure
Keywords: Control; Optimization; Heart Failure; Digital Solution
MeSH Terms: conditions — Heart Failure

STUDY DESIGN:
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (1):
- People older than 60 years with heart failure and living at home. (Experimental): People older than 60 years with heart failure and living at home.
  Interventions: Other: Digital App and Platform for Supporting Medicines Control and Optimizationin Older Individuals With Heart Failure

INTERVENTIONS:
Other: Digital App and Platform for Supporting Medicines Control and Optimizationin Older Individuals With Heart Failure — Digital App and Platform for Supporting Medicines Control and Optimizationin Older Individuals With Heart Failure

SUMMARY:
The intervention being piloted in this study is a novel system of supporting older individuals (>60 years old) with heart failure to self-manage their chronic condition through the use at home of a digital health tool that facilitates the collection and visualisation of their health data and also enables remote visualisation by health professionals. This pilot is a feasibility study in order to have a first evaluation of the engagement and user-perceived usefulness of the novel system in a real-world environment. An equivalent study will be carried out in Germany (GEWI institute). In addition, collected data will serve to validate retrospectively a heart failure decompensation prediction model (VICOMTECH, Spain) and do research into correlations with disease control (TREE TECHNOLOGY, Spain). Finally, this project is undertaken within the European project SHAPES (www.shapes2020.eu).

Older person participants (users of HUMANA GROUP services) will be asked to download the SHAPES app to their own smartphone. Medical devices - specifically, a body composition scale, a blood pressure monitor, a pulse oximeter - and a non-medical, CE-marked activity wristband, will also be provided to participants for use at home. Participants will be encouraged to take daily readings with medical devices and wear the wristband at all times. Participants can view their data via the app, which collects the readings either via Bluetooth or manually inserted by the participant. Participants will also be encouraged to complete surveys via a chatbot in the app, with questions about health status (daily), the use of medicines (weekly) and whether there are updates in medication, use of health care resources or lab test results (as required).

Health professional participants (medical doctors at HUMANA GROUP) will be able to visualise some of the collected data via: 1) eCare dashboard (data from medical devices; it is worth highlighting that they will only visualise the data coming from medical, that is not from the wristband, in order to avoid interference of non-medical information); and 2) ROSA dashboard (data from surveys and other medical data collected at baseline and during the intervention, i.e. medication, use of health care resources and lab test results). Health professional participants will use the dashboards on a daily basis and may decide to contact the older person participants for further medical evaluation.

DETAILED DESCRIPTION:
INTRODUCTION AND FINDINGS People who are aged 65 years and older account for almost a fifth of the population of the European Union. The number of people in this age group is projected to reach 151 million in 2060. Thus, there is an imperative to keep people healthy and active as they age. As age increases, however, so too does the prevalence of people living with long term conditions and subsequently, the number and complexity of treatment regimens to manage those conditions, also known as polypharmacy. In addition, the location of care delivery is also adapting - shifting routine care from hospitals to homes and the community. Home is a more comfortable and familiar setting for people and, as it has been the case during the COVID-19 pandemic, home is safer too. Individuals with chronic health conditions require regular and specialist care and support. The use of information and communication technologies (eHealth) offers opportunities to support and enhance home care.

Health literacy and individual involvement will be key elements in the successful introduction of eHealth into the health and social care system. The Smart & Healthy Ageing through People Engaging in Supportive Systems (SHAPES) Innovation Action (www.shapes2020.eu), a European project in which HUMANA GROUP is a member, intends to build, pilot and deploy a large-scale, EU-standardised open platform. SHAPES large-scale piloting campaign will engage +2k older individuals in 15 pilot sites in 10 EU Member States, including six European Innovation Partnership on Active and Healthy Ageing (EIP on AHA) Reference Sites, and involve hundreds of key stakeholders. SHAPES multidisciplinary approach to large-scale piloting is reflected across seven themes that, together, provide a clear understanding of the reality of European health and care systems and enable the validation of cost-efficient, interoperable and reliable innovations capable of effectively supporting healthy and independent living of older individuals within and outside the home.

The Medicines Optimisation Innovation Centre (MOIC), which is hosted by the Northern Health and Social Care Trust (NHSCT) is an EIP on AHA reference site and is dedicated to driving innovation in medicines use. The MOIC is leading Pilot Theme 3 of the SHAPES pilot: 'Medicines control and optimisation', wherein the SHAPES platform and selected digital solutions will be used to help participants self-monitor their health condition(s), physiological parameters and medicines adherence. Within this pilot theme there are multiple 'use cases' each deploying and evaluating different digital solutions in several European countries according to the type of support required. Four use cases will be used to evaluate this pilot theme. The project in this document describes the piloting of the use case led by CLINIKA DE KAY and carried out in Mallorca, Spain.

The use case of this project study focuses on older persons with a heart failure condition in stages 2 (patients have minor limitations while performing physical activities) or 3 (minimal ordinary activity results in weakness). Main symptom which limits quality of life is shortness of breath when patient exerts themselves or even at rest. It reduces capacity of patient to perform daily activities. An optimal management of the disease by patients is essential to prevent decompensation, a sudden functional deterioration of the heart that may lead to hospitalisation.

The combination of multiple medicines along with, many times, a change in life-style makes the management of the disease difficult. In addition, factors associated with age increase the complexity for older individuals. Adherence to treatment and life-style is usually not optimal. Finally, many individuals of this group should go to medicine reconciliation, a process which is not widely extended in health services.

The SHAPES platform along with selected digital solutions belonging to partners of the SHAPES consortium (eCare from EDGENEERING and ROSA from HUMANA GROUP) can become eHealth tools for disease self-management that are particularly designed for older persons. In addition to self-management, they provide digital complements to share data with health professionals, thus helping the integration of home disease self-management and health services. In the presented project, the main objective is to evaluate whether users engage with such a system and if it is useful for them (self-perceived usefulness).

HYPOTHESIS AND OBJECTIVES Hypothesis: This study will test the hypothesis that the SHAPES platform and Digital Solutions (novel system) are capable of providing opportunities for supporting the management of the heart failure condition, by both older persons/caregivers and health professionals.

Objectives Primary objectives

* To investigate user engagement with the novel system.
* To investigate the user-perceived usefulness of the novel system. Secondary objectives
* To investigate the capability of the novel system to optimise the use of medicines in homes:

  * Novel system triggers contacts between health professionals and patients resulting in medication change;
  * Improving medical adherence to pharmaceutical treatments.
* To investigate the capability of the novel system to improve the management of medical conditions.
* To investigate the identification of associations between precursor signs of deterioration and healthcare resource use.
* To investigate the use of Statistical Process Control (SPC) techniques to find associations between blood pressure, weight, heart rate and O2 saturation and healthcare resource use.
* To investigate the association of the VICOM's heart failure decompensation prediction score with healthcare resource use, particularly hospitalisations.
* To investigate the association of the first (active / sedentary behaviour) and second level (active in activities of daily living / intermediate activity / exercise) of physical activity classification and sleep quality analysis with healthcare resource use.
* To investigate the capability of the novel system to improve older individual's quality of life, wellbeing and psychological and psychosocial aspects.
* To explore the integration of the novel system to align with current care pathways (SO9).
* To explore user trust and acceptance of the novel system. Tertiary objectives

The following objectives align with the general purposes of the SHAPES large-scale piloting campaign:

* To validate the capability of the SHAPES Platform and Digital Solutions to support and extend healthy and independent living for older individuals who are facing permanently or temporarily reduced functionality and capabilities.
* To validate the capability of the SHAPES Platform and Digital Solutions to improve the older individuals' health outcomes and quality of life.
* To validate the capability of the SHAPES Platform and Digital Solutions to gain the older individuals' trust and acceptance.
* To validate the capability of the SHAPES Platform and Digital Solutions to gain the care professionals' trust and acceptance.
* To validate the capability of the SHAPES Platform and Digital Solutions to contribute for the reduction of the workload of medical professionals.
* To validate the capability of the SHAPES Platform and Digital Solutions to deliver efficiency gains in health and care delivery across Europe.

METHODOLOGY Materials CE-marked Medical devices: OMRON VIVA Smart Scale; OMRON M7 Intelli IT blood pressure meter; Beurer GmbH PO60 Bluetooth pulse oximeter.

CE-marked devices: Xiaomi Mi Band 3 activity wristband. Software from SHAPES partners: SHAPES platform (SHAPES consortium); eCare (EDGENEERING); ROSA (HUMANA GROUP); SHAPES app and web (combination of components from eCare, ROSA and Adilib chatbot engine from VICOMETECH); Heart failure decompensation prediction algorithm (VICOMTECH); Sleep quality and Physical intensity level and Vitals control (TREE TECHNOLOGY).

Other software: Excel, Libreoffice; Questionnaires: Those listed in outcomes.

Methods:

* Data integrity of non-CE software
* Recruitment of older persons and caregivers
* Screening: Members of the direct care team at HUMANA GROUP will screen their user lists for potentially eligible participants.
* Invitation
* Information sheets
* Consent to contact
* Eligibility confirmation
* Test in a controlled environment: 3 older person participants and 1 health professional will be invited to participate in a pre-study pilot for 1 week.
* Baseline procedures: Within 7 days before the start; For collected data.
* Intervention procedures:

All participants: On the first day, a face-to-face session with the researcher, participants will register in the SHAPES platform, devices and links will be provided and a training session will be given. The first week of the pilot will be considered a run-in period.

App users: during the pilot, the participant will be asked to record data via the SHAPES app with medical devices. They will be encouraged to take at least one measurement per device a day in the morning. Activity and sleep data is collected with CE-marked Xiaomi Mi Band 3, which will be encouraged to wear at all times. With the SHAPES app, the user can transfer data from the device to the app via Bluetooth or enter them manually. Participants will be encouraged via chatbot to answer questionnaires on a weekly and daily basis, respectively. In addition, participants will be encouraged to communicate through the chatbot in SHAPES app whether they have contacted a health professional, have new laboratory test results, have been hospitalised or their medication has changed. Independently to the scheduling of the questionnaires, the participants can answer them at any time or decide not to do so. In any case, the study will continue as the objective is to test the novel system in real world.

Health professionals: They will use the dashboards at least once on their working days to visualise data from medical devices, questionnaires collected by the chatbot and other collected medical data. If the health professional participant decides to contact the older person participant for a medical evaluation, they will self-complete a form describing the intervention. A medical doctor researcher will fill the grade of the intervention. Based on their own criteria, they may schedule survey reminders and pieces of advice to be shown in the chatbot.

* End of intervention (Within 14 days after the end of the intervention; For collected data): These data will be collected in face-to-face, one-to-one interviews or through forms to fill individually with the presence of a researcher for resolving doubts.
* Follow-up study procedures (3-month follow-up; For collected data): These data will be collected in face-to-face, one-to-one interviews or through forms to fill individually with the presence of a researcher for resolving doubts.

Data management CLINIKA DE KAY will be the data controller for all data collected during this pilot. Data Processing Agreements will be put in place between CLINIKA DE KAY and each SHAPES partner who processes data. During data collection and intervention, data processing will be pseudonymised. In analysis period, data processed by partners will be de-identified.

WORK PLAN

Research team:

* Dra. Karina Anahi Ojanguren Carreira: Medical director at HUMANA GROUP, principal investigator of the study and medical doctor researcher (PI; MD-researcher).
* Esperança Lladó Pascual, project manager and researcher at HUMANA GROUP (PM)
* Ezequiel Corredera Blanco and José María Polo, technical team at HUMANA GROUP (TT-CH)
* Researchers at VIOMTECH, TREE TECHNOLOGY.
* GEWI institute (replicating site; an equivalent study will be carried out by GEWI institute)
* National University Ireland Maynooth: Coordinator SHAPES project (Coord-SHAPES)
* Northern Health and Social Health Trust, Coordinators of Pilot Theme 3 in SHAPES (PT3-SHAPES)

ELIGIBILITY:
Inclusion Criteria:

* Users of HUMANA GROUP
* Aged 60 years old or older at the time of recruitment
* Diagnosed with heart failure at stage 2-3
* Self-reported capacity (alone or with help) to use at least 2 devices among blood pressure meter, weight scale and pulse oximeter.
* Living at home or in sheltered apartments.
* Self-reported capacity to consent
* Self-reported confident user of smartphone
* Daily access to internet
* Access to an android smartphone, with android version greater or equal to 6

Exclusion Criteria:

Not meeting the inclusion criteria

Min Age: 60 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 9 (Actual)
Dates: Start 2022-07-01 (Actual); Primary Completion 2023-01-31 (Actual); Study Completion 2023-01-31 (Actual)

PRIMARY OUTCOMES:
Timestamps of login into the novel system | 3 months
  How many times the person uses the digital solution being tested. It is expected to be used once a day.
Regarding the app, identification of pages seen, page login timestamp; page logout timestamp; measurement insertion timestamp; identification if measurement is manual or automatic | 3 months
  The processed followed by the person within the app will be analised in order to study the user experience and the potential difficulties to use the app.
Technology Acceptance Model (TAM) questionnaire | End of the use of the novel system
  The Technology Acceptance Model (TAM) is designed to measure the adoption of new technology based on customer attitudes.
Short version of User Experience Questionnaire | End of the use of the novel system
  The user experience questionnaire (UEQ) is a widely used questionnaire to measure the subjective impression of users towards the user experience of products.
Notes taken at an unstructured interview | End of the use of the novel system
  Users will be able to express any comments or suggestions other than the ones collected with the questionnaires.

CONTACTS AND LOCATIONS:
Overall Officials: Karina Anahi Ojanguren Carreira, Principal Investigator — Medical Director
Locations (1):
- Clínica Humana, Palma de Mallorca, Balearic Islands, Spain

IPD SHARING:
Plan to Share IPD: No